CLINICAL TRIAL: NCT03798197
Title: An Open-label, Single-center, Randomized, Two Period, Two Sequence Crossover Study to Characterize the Effect of Food on the Bioavailability of 30 mg Estetrol (E4) Tablet in Healthy Postmenopausal Female Volunteers
Brief Title: Effect of Food on the Bioavailability of 30 mg Estetrol (E4) Tablet in Healthy Postmenopausal Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Donesta Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MIT-Do001-C101; 2018-003761-34 (EudraCT Number)
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Food-effect
Keywords: Estetrol; Menopausal hormone therapy
MeSH Terms: interventions — Estetrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30 mg estetrol (E4) without food (fasted) (Active Comparator): Treatment A (reference): One 30 mg E4 tablet administered orally following an overnight fast of at least 10 hours.
  Interventions: Drug: 30 mg estetrol (E4)
- 30 mg estetrol (E4) with food (fed) (Experimental): Treatment B (test): One 30 mg E4 tablet administered orally 30 min after the start of an FDA prescribed high-fat breakfast preceded by at least a 10 hours overnight fast.
  Interventions: Drug: 30 mg estetrol (E4)

INTERVENTIONS:
Drug: 30 mg estetrol (E4) — All subjects received both Treatment A and Treatment B either at the first treatment period (Period 1) or at the second treatment period (Period 2). Approximately half of the subjects was randomized to receive either Treatment A followed by Treatment B (sequence AB), or Treatment B followed by Treatment A (sequence BA).
  Other Names: 30 mg E4 tablet

SUMMARY:
Assessment of the effect of a high fat meal on the quantity in blood of a female sex hormone called estetrol (E4).

The study also aims at determining how subject tolerate the study drug and how safe it is for them.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy postmenopausal females as determined by medical history, physical examination including breast examination, gynecological examination, cervical smear (Pap smear) if subject has cervix, vital signs, and laboratory tests performed within 28 days before first study drug intake.
* Between the ages of 40 and 65 years inclusive at the time of signing the informed consent (IC).
* Between the Body Mass Index (BMI) of 18 and 30 kg/m2 inclusive and body weight ≥ 45 kg.
* For non-hysterectomized women: intact uterus with bi-layer endometrial thickness ≤ 5 mm on transvaginal ultrasound (TVUS).
* Non-smokers.
* Negative test results for selected drugs of abuse and cotinine.
* Venous access sufficient to allow blood sampling as per the protocol.
* Subject is able to understand and comply with the protocol requirements, instructions, and protocol-stated restrictions.
* Subject has provided signed and dated written IC before participation in the study.

Exclusion Criteria:

* For non-hysterectomized women: uterine disease or medical condition including:

  * Bi-layer endometrial thickness >5mm as determined by TVUS;
  * Presence of fibroid(s) that obscure(s) evaluation of endometrium by TVUS;
  * History or presence of uterine cancer;
  * Presence of any significant uterine, ovarian or other adnexa related abnormality as determined by TVUS;
  * Presence of an endometrial polyp.
* Undiagnosed vaginal bleeding in the last 12 months.
* Any history of malignancy.
* History of venous or arterial thromboembolic disease
* Abnormal blood pressure.
* Use of :

  * Any prescription drugs within 28 days prior to the first study dose administration.
  * Any over-the-counter (OTC) medication or dietary supplements (vitamins included) within 14 days prior to the first study dose administration.
* Users of progestin implants or oestrogen alone injectable drug therapy are not allowed to participate unless treatment was stopped more than 3 months prior to screening.
* Users of oestrogen pellet or progestin injectable drug therapy are not allowed to participate unless treatment was stopped more than 6 months prior to screening.
* Subjects who are not in euthyroid condition.
* History of hypersensitivity or existing contraindication to E4 or intolerance to any component of the formulations or test meal.
* Presence or history of gallbladder disease, unless cholecystectomy has been performed.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the study.
* History or presence of immunodeficiency diseases including a positive human immunodeficiency virus (HIV) test result, positive hepatitis B surface antigen (HBsAg) or hepatitis C test result.
* History of illicit drug or alcohol abuse within 12 months prior to first study dose or evidence of such abuse as indicated by laboratory values within 28 days prior to first study dose.
* Consumption of foods or beverages containing the following products during the specified timeframes prior to study drug administration in Period 1: caffeine or xanthine - 48 hours; alcohol - 48 hours; grapefruit/seville orange/citrus fruit and/or star fruit - 7 days. Others Fruit juices: 72 hours prior to study drug administration.
* Donation or loss of

  * ≥ 450 mL blood within 1 month prior to initial study drug administration.
  * ≥ 250 mL blood within 2 weeks prior to initial study drug administration.
* Sponsor, Contract Research Organization (CRO) or Investigator's site personnel or their relatives directly affiliated with this study.
* History or presence of clinically relevant disease of any major system organ class (SOC) (e.g. cardiovascular, pulmonary, renal, hepatic, gastrointestinal, reproductive, endocrinological, neurological, psychiatric or orthopedic disease) as judged by the Investigator.
* Previous completion or withdrawal from this study.
* Participation in another investigational drug clinical study within 1 month (30 days) or have received an investigational drug within the last 3 months (90 days) prior to study entry.
* Is judged by the Investigator to be unsuitable for any reason.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-04-06 (Actual); Study Completion 2019-04-06 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of Estetrol in plasma | Predose, 10, 20, 30, 45 min, 1, 1.25, 1.5, 1.75, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 hours post-dose
  PK sampling
Area under the curve (AUC) from time zero to the last determinable concentration of Estetrol | Predose, 10, 20, 30, 45 min, 1, 1.25, 1.5, 1.75, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 hours post-dose
  PK sampling
AUC0-inf of Estetrol | Predose, 10, 20, 30, 45 min, 1, 1.25, 1.5, 1.75, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 hours post-dose
  PK sampling

SECONDARY OUTCOMES:
Time of Cmax (Tmax) | Predose, 10, 20, 30, 45 min, 1, 1.25, 1.5, 1.75, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 hours post-dose
  PK sampling
Terminal phase rate constant (ke) | Predose, 10, 20, 30, 45 min, 1, 1.25, 1.5, 1.75, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 hours post-dose
  PK sampling
Terminal half-life (t1/2) | Predose, 10, 20, 30, 45 min, 1, 1.25, 1.5, 1.75, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 hours post-dose
  PK sampling
Number of subjects with adverse events as measure of safety and tolerability | From Day 28 prior screening to end of study (Day 4 of Period 2)

CONTACTS AND LOCATIONS:
Overall Officials: Dobrin Svinarov, MD, Principal Investigator — MC Comac Medical Ltd.
Locations (1):
- MC Comac Medical Ltd., Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No